CLINICAL TRIAL: NCT02265822
Title: Assessment of the Effects of Melatonin on Preoperative Anxiety and Postoperative Analgesia in Children Undergoing Surgery: a Prospective, Randomized Clinical Trial
Brief Title: Melatonin Premedication in Children Undergoing Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Collaborators: Eloisa Gitto (Unknown); Lucia Marseglia (Unknown); Gabriella D'Angelo (Unknown); Sara Manti (Unknown); Simona Montalto (Unknown); Pietro Impellizzeri (Unknown)
Responsible Party: Principal Investigator, Carmelo Romeo MD, MSc, Professor, Azienda Ospedaliera Universitaria Policlinico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 797/2012
Record Dates: First submitted 2014-10-07; First posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Premedication; Anaesthesia
Keywords: melatonin; midazolam; children
MeSH Terms: interventions — Melatonin; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- melatonin (Experimental): 0.5 mg/kg (max 20 mg) oral melatonin premedication will be administered approximately 40 min before the induction of general anaesthesia with propofol. The melatonin will be prepared in a fixed volume of 5 ml adding water in a syringe without needle.
  Interventions: Drug: melatonin in children premedication
- midazolam (Active Comparator): 0.5 mg/kg (max 20 mg) oral midazolam premedication will be administered approximately 40 min before the induction of general anaesthesia with propofol. The melatonin will be prepared in a fixed volume of 5 ml adding 5% dextrose in a syringe without needle.
  Interventions: Drug: midazolam in children premedication

INTERVENTIONS:
Drug: melatonin in children premedication
  Arms: melatonin
Drug: midazolam in children premedication
  Arms: midazolam

SUMMARY:
Melatonin has been proposed as alternative to midazolam as a premedication in procedures preceding anaesthesia induction. The objective of this prospective, randomized, double-blind study is to investigate the possible effect of melatonin premedication on the required infusion of propofol in comparison to midazolam, evaluating the efficacy of oral melatonin on sedation in children undergoing surgery.

Preoperative anxiety and postoperative analgesia are also assessed in both groups.

DETAILED DESCRIPTION:
Children between the age of 5 and 14 years scheduled for elective surgery will be prospectively enrolled between September 2012 and October 2013. A physician will perform the clinical examination for each child, and anamnestic data will be collected in the medical records. Exclusion criteria will be: patients who had taken benzodiazepines, opioid drugs, or other sedative in the previous month; those who had sedation previously, or those with a temperament disorder, patients undergoing emergency surgery. Patients will be randomly assigned to 2 groups based on whether they will receive 0.2 mg/kg (max 5 mg) oral melatonin premedication (group A) or 0.5 mg/kg (max 20 mg) oral midazolam premedication (group B) before induction anaesthesia with propofol. For elective surgery, premedication will be performed between 07:30 and 09:30 h. Approximately 40 min before the induction of general anaesthesia, patients will be transported in a quiet room in the operating suite where they will receive orally melatonin or midazolam. The melatonin will be prepared by a dedicated resident in a fixed volume of 5 ml adding water in a syringe without needle. To simulate the sweet taste of the formulation of melatonin used, midazolam will be expanded to the fixed volume with 5% dextrose. The content of the syringe, in both cases marked with a coded label, will be blindly administrated to patients by the attendant nurse, not involved in the study. The child's level of sedation will be assessed and recorded by a resident before the premedication and 40 min after the administration of melatonin or midazolam, using the University of Michigan Sedation Scale (UMSS). In the operating room, an initial bolus dose of 1 mg/kg of intravenous propofol will be administered to both groups, followed by similar bolus doses of propofol until the patient will be anesthetized. Children will be considered anesthetized when asleep and not arousable. Anaesthesia will be maintained with inhalated sevoflurane. The total dose of propofol administrated will be recorded by the anaesthetist blinded to premedication group assignment. To provide objective information on the physical condition of patients after anaesthesia, Aldrete scale will be calculated after 10 min from conclusion of anaesthesia. Preoperative anxiety and postoperative analgesia will be also assessed in both groups.

ELIGIBILITY:
Inclusion Criteria:

- Children between the age of 5 and 14 years scheduled for elective surgery

Exclusion Criteria:

* Patients who had taken benzodiazepines, opioid drugs, or other sedative in the previous month
* Those who had sedation previously, or those with a temperament disorder, patients undergoing emergency surgery

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
efficacy of melatonin as premedicant in children undergoing elective surgery | day 1: 40-45 min after melatonin or midazolam premedication
  the required infusion of propofol required during induction of general anaesthesia in both groups will be evaluated

SECONDARY OUTCOMES:
effect of melatonin premedication in postoperative analgesia in children undergoing elective surgery | day 1: 40 min after melatonin or midazolam premedication
  The child's level of sedation will be assessed and recorded using the University of Michigan Sedation Scale (UMSS).
effect of melatonin premedication in postoperative analgesia in children undergoing elective surgery | day 1: 3, 6, and 12 hours post surgery
  post procedural pain will be assessed and recorded in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Romeo, Prof, Study Chair — Azienda Ospedaliera Universitaria Policlinico "G. Martino"

REFERENCES:
- [Result] Acil M, Basgul E, Celiker V, Karagoz AH, Demir B, Aypar U. Perioperative effects of melatonin and midazolam premedication on sedation, orientation, anxiety scores and psychomotor performance. Eur J Anaesthesiol. 2004 Jul;21(7):553-7. doi: 10.1017/s0265021504007094. PMID 15318468
- [Result] Naguib M, Gottumukkala V, Goldstein PA. Melatonin and anesthesia: a clinical perspective. J Pineal Res. 2007 Jan;42(1):12-21. doi: 10.1111/j.1600-079X.2006.00384.x. PMID 17198534
- [Result] Naguib M, Samarkandi AH, Moniem MA, Mansour Eel-D, Alshaer AA, Al-Ayyaf HA, Fadin A, Alharby SW. The effects of melatonin premedication on propofol and thiopental induction dose-response curves: a prospective, randomized, double-blind study. Anesth Analg. 2006 Dec;103(6):1448-52. doi: 10.1213/01.ane.0000244534.24216.3a. PMID 17122221
- [Result] Kurdi MS, Patel T. The role of melatonin in anaesthesia and critical care. Indian J Anaesth. 2013 Mar;57(2):137-44. doi: 10.4103/0019-5049.111837. PMID 23825812